CLINICAL TRIAL: NCT06378151
Title: Time-limited Trials in the Emergency Department: A Randomized Trial
Brief Title: Time-limited Trials in the Emergency Department
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Kei Ouchi, Associate Professor of Emergency Medicine, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2023P002243
Record Dates: First submitted 2024-02-08; First posted 2024-04-22 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Emergencies
Keywords: Time-Limited Trials; emergency department; palliative care
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Intervention Model Description: Clinician-level randomization
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): Attending physicians, resident physicians, or mid-level providers working in the ED who are willing to be randomized to become the study interventionists.
  Interventions: Other: TLT training
- Control group (No Intervention): Attending physicians, resident physicians, or mid-level providers working in the ED who are willing to be randomized to become the study interventionists.

INTERVENTIONS:
Other: TLT training — Emergency clinicians assigned to the intervention group will receive the following training and resources.
  1. The TLT Conversation Guide: The structured conversation guide entails discussing patients' values and goals, prognosis, and shared decision-making to use a trial of intensive care. Originally used in ICU settings, we systematically refined the guide to be used in the ED incorporating inputs from patient advisors' and emergency clinicians' inputs.
  2. Clinician Training: The clinician training will include a one-hour didactic on research methodologies and serious illness communication skills, followed by a four-hour communication training with trained actors.
  3. EHR Documentation: An EHR template for documenting the TLT conversation findings has been developed.
  4. Intensivist Communication: A standard template to communicate the TLT conversation findings to the intensivists has been developed.
  Arms: Intervention group

SUMMARY:
A randomized controlled trial of a structured conversation between clinicians and patients/surrogates to facilitate shared decision-making for intensive care use in seriously ill older adults being admitted to the intensive care unit from the emergency department.

DETAILED DESCRIPTION:
A randomized controlled trial of a structured conversation between clinicians and patients/surrogates to facilitate shared decision-making for intensive care use (i.e., Time-Limited Trial, TLT) in seriously ill older adults being admitted to the intensive care unit from the emergency department (ED).

The goal is to evaluate the feasibility and acceptability of TLT initiated in the ED for seriously ill older adults who are starting intensive care.

The main questions it aims to answer are:

* Is TLT feasible to be conducted by trained ED clinicians?
* Do patients or their surrogates find TLT acceptable in understanding and respecting their end-of-life care preferences?

Participants will be:

* Attending physicians, resident physicians, or mid-level providers working in the ED who are willing to be randomized to become the study interventionists to conduct TLT conversations.
* Seriously ill older adults receiving intensive care in the ED.

Researchers will compare clinicians using TLT with those providing usual care to see if TLT leads to improved patient-centered decision-making and better alignment with patients' end-of-life care preferences.

ELIGIBILITY:
Physician's eligibility:

Inclusion Criteria:

* Attending physicians, resident physicians, or mid-level providers working in the ED who are willing to be randomized to become the study interventionists.

Exclusion Criteria:

* Emergency clinicians unwilling to consent and be randomized to intervention TLT training.

Patient's eligibility:

The subjects will be seriously ill older adults, or their surrogates being cared for by the participating emergency clinicians (both the intervention or control arms). If the emergency clinicians determine that the patient is not able to provide consent due to cognitive impairment, dementia, delirium, or critical illness, the surrogates will participate in the TLT conversations.

Inclusion Criteria:

1. ≥50 years or older with ≥one serious life-limiting illness* being admitted to the intensive care unit in the ED; or
2. ≥75 years or older being admitted to intensive care unit in the ED; or
3. ED clinicians will not be surprised if the patient died in the current hospital admission or in the near future; and
4. English speaking *Serious illness criteria with high one-year mortality are selected based on best practice recommendations such as 1) stage III/IV or metastatic cancer; 2) end-stage renal disease on dialysis; 3) chronic heart/lung disease requiring home oxygen supplementation or experiencing shortness of breath with walking; 4) moderate to severe dementia (surrogate required for enrollment); or 5) ≥2 hospitalizations or ED visits in the past six months.

Exclusion Criteria:

1. Unable or unwilling to provide informed consent; or
2. Non-English speaking; or
3. Clinically inappropriate, determined by emergency clinicians, and no surrogate is available

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-04-12 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Time to complete TLT conversations | Immediately after the intervention (TLT conversation)
  With direct observation, the study team will record how long (e.g., minutes) it takes to complete the TLT conversations by the interventionist ED clinicians.
Patient-reported acceptability of TLT conversations | Immediately after the intervention (TLT conversation)
  A 5-point Likert scale (i.e., "How acceptable was it for your doctor to talk to you about your expectations for ICU care?" and "How likely would you recommend this conversation for other patients like you?" "Not at all (1)" to "Completely (5)"). A higher score indicates a better outcome.

SECONDARY OUTCOMES:
Intervention fidelity | Immediately after the intervention (TLT conversation)
  With direct observation, the study team will record the completion of TLT components using an intervention fidelity checklist.
Clinician-reported feasibility | Immediately after the intervention (TLT conversation)
  The study team will ask the interventionist emergency clinician to complete two 5-point Likert scale questions. The scale includes the following response options: "not at all (1)," "slightly (2)," "moderately (3)," "quite a bit (4)," and "completely (5)." A higher score indicates a better outcome.
Clinician-reported satisfaction | Immediately after the intervention (TLT conversation)
  The study team will ask the interventionist emergency clinician to complete 5-point Likert scale questions (i.e., "How satisfied are you with the conversation? "Not at all (1)," "slightly (2)," "moderately (3)," "quite a bit (4)," and "completely (5)"). A higher score indicates a better outcome.
Clinician-reported likelihood of recovery | At enrollment
  A 5-point Likert scale to identify clinicians' reported likelihood of their patient's recovery to their baseline function regarding the patient's quality of life, physical function, and cognitive function. The scale includes the following response options: "very unlikely (1)," "unlikely (2)," "neutral / neither likely nor unlikely (3)," "likely (4)," and "very likely (5)." Higher scores indicate a greater clinician-reported likelihood of recovery.
EHR documentation by inpatient clinicians | After 24 hours, 48 hours, and 1 week
  Review EHR for new documentation of reference to TLT, serious illness conversation, change in code status, or advance directive forms by inpatient clinicians.
Heard and understood | Immediately after the intervention (TLT conversation)
  A National Quality Forum endorsed, validated measure for palliative care modified to fit the context of serious illness conversations. This instrument is a 5-point Likert scale: "not at all (1)," "slightly (2)," "moderately (3)," "quite a bit (4)," and "completely (5)." A higher score indicates a better outcome.
Patient-reported end-of-life quality of communication | Immediately after the intervention (TLT conversation)
  A validated, quality of end-of-life communication survey. This instrument is a 10-point Likert scale ranging from "the very worst I could imagine (0)" to "the very best I could imagine (10)". A higher score indicates a better outcome.
Patient-reported likelihood of recovery | At enrollment
  A 5-point Likert scale to identify patients'/surrogates' understanding of the likelihood of the patient's recovery to their baseline function regarding their quality of life, physical function, and cognitive function. The scale includes the following response options: "very unlikely (1)," "unlikely (2)," "neutral / neither likely nor unlikely (3)," "likely (4)," and "very likely (5)." Higher scores indicate a greater patient-reported likelihood of recovery.
Needs at the end-of-life screening tool | At enrollment, after 24 hours, after 48 hours, and after 1 week
  Two questions from a validated, survey (Needs at the End-of-life Screening Tool) on the clarity of the information provided by the clinician, and on the patient's goals of care. This instrument is a 10-point Likert scale ranging from "not at all (0)" to "completely (10)". A higher score indicates a better outcome.
Patient-reported anxiety scale | At enrollment, after 48 hours, and after 1 week
  A subscale of the validated Hospital Anxiety and Depression Scale (HADS), the HADS-Anxiety (HADS-A) subscale will be used to assess patients' or surrogates' anxiety levels. Scores range from 0 to 21, with higher scores indicating greater anxiety.
Decisional regret scale | After 24 hours, 48 hours, and 1 week
  A five-item validated survey of decisional regret. This instrument is a 5-point Likert scale: "strongly agree (1)," "agree (2)," "neither agree nor disagree (3)," "disagree (4)," and "strongly disagree (5)." The results will be converted into a score from 0 to 100. A higher score indicates greater regret.
The number of days to the first family meeting in ICU | Immediately after patient's discharge or death
  The number of days from ICU admission to the first family meeting was documented by the ICU clinical team.
ICU length of stay (LOS) | Immediately after patient's discharge or death
  The ICU LOS is recorded in days, from admission to the ICU until discharge, based on hospital records.
Hospital LOS | Immediately after patient's discharge or death
  Hospital LOS is recorded in days, from admission to the hospital until discharge, as recorded in the patient's hospital record.
The number of family meetings | Immediately after patient's discharge or death
  The total number of family meetings conducted in the ICU, as documented in patient records.
ICU procedures (e.g., CPR, pressors, etc.) | Immediately after patient's discharge or death
  The number and type of specific ICU procedures performed, such as CPR or the use of pressors, will be recorded for each patient.
ICU mortality | Immediately after patient's discharge or death
  ICU mortality is the percentage of patients who die while in the ICU, documented by the hospital's patient management system.
Patterns of hospital disposition | Immediately after patient's discharge or death
  Hospital disposition refers to the patient's status upon discharge, including return home, transfer to another facility, or death, as noted in discharge records.
Rate of hospice utilization | Immediately after patient's discharge or death
  Hospice utilization is recorded as the incidence of patients transferred to hospice care from the hospital, verified by hospice admission records.

CONTACTS AND LOCATIONS:
Overall Officials: Kei Ouchi, MD, MPH, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gramling R, Stanek S, Ladwig S, Gajary-Coots E, Cimino J, Anderson W, Norton SA; AAHPM Research Committee Writing Group; Aslakson RA, Ast K, Elk R, Garner KK, Gramling R, Grudzen C, Kamal AH, Lamba S, LeBlanc TW, Rhodes RL, Roeland E, Schulman-Green D, Unroe KT. Feeling Heard and Understood: A Patient-Reported Quality Measure for the Inpatient Palliative Care Setting. J Pain Symptom Manage. 2016 Feb;51(2):150-4. doi: 10.1016/j.jpainsymman.2015.10.018. Epub 2015 Nov 17. PMID 26596879
- [Background] Engelberg R, Downey L, Curtis JR. Psychometric characteristics of a quality of communication questionnaire assessing communication about end-of-life care. J Palliat Med. 2006 Oct;9(5):1086-98. doi: 10.1089/jpm.2006.9.1086. PMID 17040146
- [Background] Brehaut JC, O'Connor AM, Wood TJ, Hack TF, Siminoff L, Gordon E, Feldman-Stewart D. Validation of a decision regret scale. Med Decis Making. 2003 Jul-Aug;23(4):281-92. doi: 10.1177/0272989X03256005. PMID 12926578
- [Derived] Hashimoto T, Putman RK, Massaro AF, Shiozawa Y, McGough K, McCabe KK, Linden JA, Wang W, Liu SW, Kennedy M, Neville TH, Kruser JM, Sudore RL, Schonberg MA, Tulsky JA, Ouchi K. Study protocol for a randomized controlled trial: Integrating the 'Time-limited Trial' in the emergency department. PLoS One. 2024 Dec 23;19(12):e0313858. doi: 10.1371/journal.pone.0313858. eCollection 2024. PMID 39715103